CLINICAL TRIAL: NCT07083817
Title: A Single-dose, Phase 1, Open-label Study to Evaluate the Mass Balance and Absorption, Distribution, Metabolism, and Excretion of [14C]Xeruborbactam (QPX7728) Following Administration of a Solution for Intravenous Infusion in Healthy Adult Male Participants
Brief Title: Mass Balance Study of [14C]Xeruborbactam (QPX7728) in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qpex Biopharma, Inc. (Industry)
Collaborators: Shionogi Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Qpex-403
Record Dates: First submitted 2025-07-11; First posted 2025-07-24 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: ADME

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C]Xeruborbactam (Experimental)
  Interventions: Drug: [14C]Xeruborbactam

INTERVENTIONS:
Drug: [14C]Xeruborbactam — Carbon Radiolabeled Xeruborbactam

SUMMARY:
This is a single-dose, phase 1 open-label study to determine the mass balance recovery and metabolic profiling and identification for intravenous (IV) administered [14C]xeruborbactam. This study will investigate the primary route of excretion, profile [14C]xeruborbactam metabolites in plasma, urine and faeces, and assess the safety, tolerability, and pharmacokinetics (PK) of a single IV dose of [14C]xeruborbactam in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, safety laboratory tests, vital signs, and cardiac (12-lead electrocardiogram (ECG)) monitoring.
* Body weight within 55.0 and 100.0 kg (inclusive) and body mass index (BMI) within the range of 18.0 and 32.0 kg/m2 (inclusive).
* Participants who have regular bowel movements (ie, average stool production of ≥ 1 and ≤ 3 stools per day)
* Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent

Exclusion Criteria:

* History or presence of significant cardiovascular, respiratory/pulmonary, hepatic, renal, hematological, gastrointestinal (GI), endocrine, immunologic, dermatologic, neurological, or psychiatric disease capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the investigational intervention; or interfering with the interpretation of data
* Surgery within the past 3 months prior to Day 1 determined by the investigator to be clinically relevant
* History of GI surgery including but not limited to, gastric resection and/or intestinal resection that may result in a clinically significant abnormality in GI function (expect for an appendectomy for noncomplicated appendicitis unless it was performed in the previous 12 months)
* Acute diarrhea, loose stools, or constipation within 14 days prior to the screening visit or upon admission to the clinical research unit (CRU) (Day -1). Diarrhea will be defined as the passage of liquid faeces and/or a stool frequency of ≥ 3 times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-08-13 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Amount of total radioactivity excreted expressed as a percentage of the radioactive dose administered (Fe) | Day 1 to Day 15
Cumulative amount of total radioactivity excreted expressed as percentage of the radioactive dose administered (CumFe) | Day 1 to Day 15
Ratio of plasma xeruborbactam concentrations relative to total radioactivity based on Cmax | Day 1 to Day 15
Ratio of plasma xeruborbactam concentrations relative to total radioactivity based on AUC0-last | Day 1 to Day 15
Ratio of plasma xeruborbactam concentrations relative to total radioactivity based on AUC0-inf | Day 1 to Day 15
Whole blood to plasma total radioactivity ratio based on Cmax | Day 1 to Day 15
Whole blood to plasma total radioactivity ratio based on AUC0-last | Day 1 to Day 15
Whole blood to plasma total radioactivity ratio based on AUC0-inf | Day 1 to Day 15
Maximum plasma concentration (Cmax) for xeruborbactam | Day 1 to Day 15
Time to maximum plasma concentration (Tmax) for xeruborbactam | Day 1 to Day 15
Area under the concentration time curve from zero to infinity (AUC0-inf) for xeruborbactam | Day 1 to Day 15
Maximum plasma and whole blood concentration (Cmax) of total radioactivity | Day 1 to Day 15
Time to maximum plasma and whole blood concentration (Tmax) of total radioactivity | Day 1 to Day 15
Area under the concentration time curve from zero to infinity (AUC0-inf) of total radioactivity in plasma and whole blood | Day 1 to Day 15
Amount of total radioactivity excreted in urine (Aeu) | Day 1 to Day 15
Amount of total radioactivity excreted in in urine expressed as a percentage of the radioactive dose administered (Feu) | Day 1 to Day 15
Identification of the chemical structure of each metabolite accounting for 5% or more in plasma by area under the time concentration curve (AUC) | Day 1 to Day 15
Identification of the chemical structure of each metabolite in urine and faeces that account for 5% or more of the administered radioactive dose | Day 1 to Day 15
Total amount of radioactivity excreted (Ae) | Day 1 to Day 15
Cumulative amount of total radioactivity excreted (CumAe) | Day 1 to Day 15
Ratio of whole blood to plasma total radioactivity | Day 1 to Day 15

SECONDARY OUTCOMES:
Percentage of participants with Treatment-Emergent Adverse Events | Day 1 to Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom